CLINICAL TRIAL: NCT05328154
Title: Effects of the Combination of Magnesium Bisphosphonates Versus Bisphosphonates Alone on Bone Remodeling: Randomized Pilot Clinical Trial
Brief Title: MAGnesium Effect With ANtiosteoporotic Drugs
Acronym: MAGELLAN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AOI 2021 ME_PICKERING; 2021-005401-28 (EudraCT Number)
Record Dates: First submitted 2022-03-29; First posted 2022-04-14 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Osteoporosis, Postmenopausal
Keywords: Osteoporosis; Magnesium; CTX; Bone remodeling
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis | interventions — Nuclear Receptor Subfamily 4, Group A, Member 2

STUDY DESIGN:
Intervention Model Description: Following the inclusion visit, patients will be assigned to one of the two groups (bisphosphonates alone or bisphosphonate associated with magnesium). Treatment assignment will follow a predefined randomization list and will be performed by a Clinical Research Associate who is totally independent from the protocol. The randomization list and a copy will be edited and given to the Clermont-Ferrand University Hospital Pharmacy and to the Rheumatology Department of the Gabriel Montpied University Hospital.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bisphosphonates (zoledronic acid, Aclasta® 5 mg) alone (Other): Bisphosphonates are considered as the gold standard of treatment for osteoporosis. Zoledronic acid, Aclasta® 5 mg will be administered intravenously according to standard management criteria in order to obtain an homogeneous population.
  Interventions: Other: Follow-up of patients with postmenopausal osteoporosis, with or without fractures, requiring initiation of injectable bisphosphonate therapy as part of their usual care
- bisphosphonates (zoledronic acid, Aclasta® 5 mg) associated with magnesium (MAG 2®, 100 mg) (Active Comparator): In addition to bisphosphonates, patients in this group will take a 3-month treatment of magnesium (magnesium carbonate, MAG 2® 100 mg), 2 tablets of 100 mg/day, during the 3 months preceding the 1-year visit.
  Interventions: Drug: Follow-up of patients with postmenopausal osteoporosis, fractured or not, requiring initiation of injectable bisphosphonate therapy as part of care with magnesium supplementation

INTERVENTIONS:
Other: Follow-up of patients with postmenopausal osteoporosis, with or without fractures, requiring initiation of injectable bisphosphonate therapy as part of their usual care — * Inclusion medical consultation
  * Inclusion clinical examination
  * Calculation of Kauppila score at one year
  * Imaging procedures (DXA) at 1 year
  * Magnesium dosage: Visit 1: Day 0 and Visit 3: Day 0+1 year
  * Samples for biological collection and microbiota analysis Visit 1: Day 0 and Visit 3: Day 0+1 year
  * Genotyping in Visit 1: Day 0
  * Serum CTX dosage in Visit 3: Day 0+1 year
  * Cardiovascular investigations (FMD, RHI, FLD, PWV) in Visit 1: Day 0 and Visit 3: Day 0+1 year
  * Exploration of sarcopenia (SARC-F, SPPB, muscle strength and body composition) in Visit 1: Day 0 and Visit 3: Day 0+1 year
  * Exploration of pain (NPS, BPI, sensitivity/pain thresholds, CPM) in Visit 1: Day 0 and Visit 3: Day 0+1 year
  * Quality of life component questionnaires (PSQI, HADs, SF-36) in Visit 1: Day 0 and Visit 3: Day 0+1 year
  * Follow-up diary to be completed at months 1 and 12 of the study
  Arms: Bisphosphonates (zoledronic acid, Aclasta® 5 mg) alone
Drug: Follow-up of patients with postmenopausal osteoporosis, fractured or not, requiring initiation of injectable bisphosphonate therapy as part of care with magnesium supplementation — * Inclusion medical consultation
  * Inclusion clinical examination
  * Calculation of Kauppila score at one year
  * Imaging procedures (DXA) at 1 year
  * Magnesium dosage: Visit 1: Day 0; Visit 2: Day 0+9 months and Visit 3: Day 0+1 year
  * Samples for biological collection and microbiota analysis Visit 1: Day 0 and Visit 3: Day 0+1 year
  * Genotyping in Visit 1: Day 0
  * Serum CTX dosage in Visit 3: Day 0+1 year
  * Cardiovascular investigations (FMD, RHI, FLD, PWV) in Visit 1: Day 0 and Visit 3: Day 0+1 year
  * Exploration of sarcopenia (SARC-F, SPPB, muscle strength and body composition) in Visit 1: Day 0 and Visit 3: Day 0+1 year
  * Exploration of pain (NPS, BPI, sensitivity/pain thresholds, CPM) in Visit 1: Day 0 and Visit 3: Day 0+1 year
  * Quality of life component questionnaires (PSQI, HADs, SF-36) in Visit 1: Day 0 and Visit 3: Day 0+1 year
  * Magnesium intake for 1 period of 3 months
  * Phone call
  * Follow-up diary to be completed at months 1, 10, 11 and 12 of the study
  Arms: bisphosphonates (zoledronic acid, Aclasta® 5 mg) associated with magnesium (MAG 2®, 100 mg)

SUMMARY:
Randomized pilot clinical trial to demonstrate superiority of bisphosphonate-magnesium combination over bisphosphonates alone in postmenopausal osteoporosis in slowing bone remodeling as assessed by C-terminal telopeptide of bone collagen type 1 (CTX) dosage.

DETAILED DESCRIPTION:
A pilot, randomized, controlled, open-label, single-center, two-parallel-arm clinical trial testing the addition of oral magnesium supplementation to prescribed drug therapy in the care setting. Category 1.

The primary objective of this randomized trial is to demonstrate the superiority of the combination of bisphosphonates and magnesium over bisphosphonates alone in postmenopausal osteoporosis, in terms of slowing bone remodeling, as assessed by the measurement of C-terminal telopeptides of type 1 bone collagen (CTX).

The secondary objectives are to study the impact of magnesium supplementation at 1 year on:

1. the evolution of other biological markers of bone remodeling (by creating a collection of biological samples) and bone densitometry on the following sites: spine, femoral neck, total femur,
2. the evolution of cardiovascular parameters,
3. the follow-up of the incidence of fractures,
4. the evolution of sarcopenia,
5. the evolution of quality of life and pain,
6. the genetic predisposition of osteoporosis including the confirmation of known genetic markers and the potential identification of new genetic variants involved (by creating a biobank),
7. the epigenetic biomarkers in the osteoporosis patient population (by creating a biobank),
8. the role of the microbiota in osteoporosis patients (by creating a biobank),
9. the occurrence of adverse events.

As part of their usual care and management, patients will be diagnosed with osteoporosis and prescribed bisphosphonates.

Patients will have 3 or 4 visits depending on which group they are randomized to: a first screening visit as part of routine care, which will take place in the Rheumatology Department of the Clermont-Ferrand University Hospital, then 2 visits for patients in the "bisphosphonates alone" group and 3 visits for patients in the "bisphosphonates associated with magnesium" group, which will take place in the Inserm 1405 Clinical Investigation Platform/Clinical Investigation Center (PIC/CIC) of the Clermont-Ferrand University Hospital.

Visit 0 - Screening visit and diagnosis of osteoporosis (1 month before day 0): Rheumatology Department

During this visit, the investigator physician will perform various examinations and tests usually performed as part of the patient's usual care and management in order to establish a diagnosis of osteoporosis.

These examinations are as follow:

* Bone densitometry less than one year using Dual X-ray Absorptiometry (DXA), either previously performed by the patient or prescribed at this consultation.
* Bone biological assessment, including the following tests: Complete Blood Count (CBC), platelets, C-Reactive Protein (CRP), urea, creatinine with CKD-EPI clearance calculation, liver enzymes (AST, ALT), serum calcium, serum calcium corrected by albumin, serum phosphorus, serum protein electrophoresis, Thyroid Stimulating Hormone (TSH), 25 OH vitamin D, serum CTX.

Some patients who require profile radiographs of the spine will have this examination added for the consultation, especially for the evaluation of vertebral fractures if the context justifies it. Other patients will also have these x-rays to calculate the abdominal aortic calcification score (Kauppila score).

Body composition will be requested during the bone densitometry evaluation on the DXA machine.

Once the diagnosis of osteoporosis is confirmed, the physician will propose to eligible patients to participate in this research protocol by explaining the objectives and the course of the study, and give them an information note.

If the patients are interested, the investigator physician will prescribe osteoporotic treatment to be started after the Visit 1: Day 0 inclusion visit.

Visit 1 - Inclusion visit (Day 0): PIC/CIC (2 hours)

During this visit, the physician will explain again the objectives and progress of the study with the different tests and questionnaires planned so that the patients can give their informed consent to participate.

During this visit, the following will be performed:

* A medical examination,
* A blood sample to measure magnesium levels and to obtain a collection of biological samples in order to:

  1. Evaluate bone biomarkers (osteocalcin, sclerostin, periostin, irisin, N-terminal propeptide of procollagen type 1 (P1NP), Dickkopf-related protein 1 (DKK1)),
  2. Characterize genetic predispositions of osteoporosis,
  3. Characterize epigenetic biomarkers in the osteoporosis patient population by microRNA analysis,
* A stool sample to obtain a biobank for subsequent microbiota analysis.
* A cardiovascular exploration based on the measurement of the increase in the diameter of the brachial artery (FMD, "Flow-Mediated Dilation"); measurement of the increase in digital volume (RHI, "Reactive Hyperemia Index") and measurement of the microcirculatory perfusion of the skin at the level of the hand (FLD, "Flow Laser Doppler"), and measurement of the stiffness of the main arteries (aorta) by the technique of Pulse Wave Velocity (PWV) measurement.
* Exploration of sarcopenia: the following questionnaires and tests will be performed: SARC-F (Strength, Assistance with walking, Rising from a chair, Climbing stars, and Falls), SPPB (Short Physical Performance Battery), the measurement of the muscular function and DXA with the measurement of the body composition.
* Pain exploration: Numerical Pain Scale (NPS), Brief Pain Inventory (BPI), and pain thresholds.
* Quality of life component questionnaires: Pittsburgh Sleep Quality Index (PSQI), the Hospital Anxiety and Depression scale (HADs) and the 36-Item Short Form Survey (SF-36).
* Randomization into two groups: a "bisphosphonates associated with magnesium" group, and a "bisphosphonates alone" group.
* Delivery of a daily follow-up diary to evaluate the average pain per day, the consumption of analgesics, and the occurrence of any adverse effects.

For the "bisphosphonates alone" group, this diary will be completed for the first month of taking bisphosphonates (Month 1) as well as for the last month before the end of study visit at one year (Month 12).

For the "bisphosphonates combined with magnesium" group, a diary will also be given to them for the first month of taking bisphosphonates and a second will be given to them at visit 2 which will cover the period of taking magnesium over the last 3 months preceding the end-of-study visit (Months 10 to 12).

Visit 2 only for patients in the bisphosphonate-magnesium arm (Day 0+9 months): PIC/CIC (15 minutes)

At this visit, 9 months after the start of the trial, a blood test will be performed to measure magnesium levels, and then patients will be given magnesium treatment to take daily for 3 months before their 1-year visit (during months 10, 11 and 12). Finally, they will be given a follow-up diary to evaluate the average pain per Numerical Pain Scale, the daily consumption of analgesics, and the occurrence of possible adverse effects.

→ In addition, for the patients in this group, a phone call will be made by the project team 6 weeks after the start of the magnesium treatment to ensure good tolerance and compliance with the magnesium intake.

Visit 3 - End of study visit at 1 year (Day 0+1 year): PIC/CIC (1h15)

During this visit, the following examinations, tests and questionnaires will be performed:

* A medical examination,
* A blood sample to measure magnesium levels, serum CTX and other biological bone markers (osteocalcin, sclerostin, periostin, irisin, P1NP, DKK1) and to perform microRNA analysis by collecting biological samples,
* A stool sample to study the microbiota (constitution of a collection of biological samples),
* A bone densitometry measurement (DXA),
* A cardiovascular exploration with FMD, RHI, FLD and PWV measurements and an estimation of the Kauppila score.
* Exploration of sarcopenia: questionnaires and tests SARC-F, SPPB, measurement of muscle function and body composition.
* Exploration of pain: NPS, BPI, and pain thresholds.
* Quality of life component questionnaires: PSQI, HADs and the SF-36. As part of routine care, patients will then be seen in a follow-up rheumatology consultation to confirm the indication for continuing treatment with biphosphonates, with a blood test identical to that performed during the pre-selection visit.

Visit 3 will be the last visit of the study.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 50 years or older, with postmenopausal osteoporosis, fractured or not, requiring initiation of injectable bisphosphonate therapy as part of their care.
* Able to give informed consent to participate in the research.
* Affiliation to a Social Security system.

Exclusion Criteria:

* Initial densitometry more than one year old.
* Patient receiving a treatment or food supplement containing magnesium (Mg).
* Contra-indication to the administration of Mg: hypersensitivity to magnesium carbonate or to one of the excipients.
* Patients with a magnesium level > 1.07 mmol/l.
* Patient with chronic renal failure, defined as creatinine clearance < 35 mL/min estimated by Cockcroft-Gault or glomerular filtration rate < 30 mL.min-1 estimated by CKD-EPI and taking into account which is more pejorative.
* Patient with a medical and/or surgical history deemed by the investigator or his representative to be incompatible with the trial.
* Patient under legal protection or deprived of liberty.
* Refusal to participate.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
C-terminal telopeptides of collagen type 1 (CTX) dosage | Visit 0: Day 0-1 month
  Evaluation of the CTX evolution after one year, defined as the difference [after - before], relative to the basal value (ng/ml). For this purpose, a blood sample will be taken using 5 mL dry tubes.
C-terminal telopeptides of collagen type 1 (CTX) dosage | Visit 3: Day 0+1 year
  Evaluation of the CTX evolution after one year, defined as the difference [after - before], relative to the basal value (ng/ml). For this purpose, a blood sample will be taken using 5 mL dry tubes.

SECONDARY OUTCOMES:
N-terminal propeptide of procollagen type 1 (P1NP) dosage | Visit 1: Day 0
  The dosage of N-terminal propeptide of procollagen type 1 (P1NP) (µg/l) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes.
N-terminal propeptide of procollagen type 1 (P1NP) dosage | Visit 3: Day 0+1 year
  The dosage of N-terminal propeptide of procollagen type 1 (P1NP) (µg/l) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes.
Osteocalcin dosage | Visit 1: Day 0
  The dosage of osteocalcin (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes
Osteocalcin dosage | Visit 3: Day 0+1 year
  The dosage of osteocalcin (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes
Sclerostin dosage | Visit 1: Day 0
  The dosage of slerostin (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes.
Sclerostin dosage | Visit 3: Day 0+1 year
  The dosage of slerostin (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes.
Periostin dosage | Visit 1: Day 0
  The dosage of periostin (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes.
Periostin dosage | Visit 3: Day 0+1 year
  The dosage of periostin (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes.
Irisin dosage | Visit 1: Day 0
  The dosage of irisin (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken on 4 mL heparin tube for irisin dosage.
Irisin dosage | Visit 3: Day 0+1 year
  The dosage of irisin (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken on 4 mL heparin tube for irisin dosage.
Dickkopf-related protein 1 (DKK1) dosage | Visit 1: Day 0
  The dosage of Dickkopf-related protein 1 (DKK1) (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes.
Dickkopf-related protein 1 (DKK1) dosage | Visit 3: Day 0+1 year
  The dosage of Dickkopf-related protein 1 (DKK1) (ng/ml) will be performed in order to evaluate bone remodeling. For this purpose, a blood sample will be taken using 5 mL dry tubes.
Magnesium (Mg) dosage | Visit 1: Day 0
  A blood sample will be taken using 3 mL lithium heparin tube for the dosage of the magnesium (mmol/L).
Magnesium (Mg) dosage | Visit 2: Day 0+9 months
  A blood sample will be taken using 3 mL lithium heparin tube for the dosage of the magnesium (mmol/L).
Magnesium (Mg) dosage | Visit 3: Day 0+1 year
  A blood sample will be taken using 3 mL lithium heparin tube for the dosage of the magnesium (mmol/L).
Evaluation of bone densitometric parameters (femoral neck) | Visit 0: Day 0-1 month
  Densitometry analysis on the three usual sites (femoral neck) by Dual X-ray Absorptiometry (DXA). T-scores will be analyzed at these sites, as well as densitometry in grams per square centimeter.
Evaluation of bone densitometric parameters (femoral neck) | Visit 3: Day 0+1 year
  Densitometry analysis on the three usual sites (femoral neck) by Dual X-ray Absorptiometry (DXA). T-scores will be analyzed at these sites, as well as densitometry in grams per square centimeter.
Evaluation of bone densitometric parameters (total femur) | Visit 0: Day 0-1 month
  Densitometry analysis on the three usual sites (total femur) by Dual X-ray Absorptiometry (DXA). T-scores will be analyzed at these sites, as well as densitometry in grams per square centimeter.
Evaluation of bone densitometric parameters (total femur) | Visit 3: Day 0+1 year
  Densitometry analysis on the three usual sites (total femur) by Dual X-ray Absorptiometry (DXA). T-scores will be analyzed at these sites, as well as densitometry in grams per square centimeter.
Evaluation of bone densitometric parameters (spine) | Visit 0: Day 0-1 month
  Densitometry analysis on the three usual sites (spine) by Dual X-ray Absorptiometry (DXA). T-scores will be analyzed at these sites, as well as densitometry in grams per square centimeter.
Evaluation of bone densitometric parameters (spine) | Visit 3: Day 0+1 year
  Densitometry analysis on the three usual sites (spine) by Dual X-ray Absorptiometry (DXA). T-scores will be analyzed at these sites, as well as densitometry in grams per square centimeter.
Endothelial dysfunction measured by FMD (Flow-Mediated Dilation) | Visit 1: Day 0
  FMD is a non-invasive technique. It was assessed using an ultrasound approach with a high-resolution linear array transducer coupled with computer-assisted analysis software. With this software, changes in the brachial artery could be assessed in real-time through an automated edge detection system. Longitudinal images of the brachial artery were obtained with the transducer fixed on the medial aspect of the dominant arm, approximately 2 cm above the medial epicondyle of the humerus. The transducer was fixed on the arm by a special arm-holding device. The brachial artery diameter was acquired as per a 30 s baseline measure, after which a cuff was placed around forearm (3 cm above wrist) and inflated to 250 mm Hg for 5 min. After cuff deflation, the brachial artery diameter was continuously monitored for 2-4 min to detect the peak artery diameter. FMD was determined as the percentage change in diameter from baseline to peak arterial diameter.
Endothelial dysfunction measured by FMD (Flow-Mediated Dilation) | Visit 3: Day 0+1 year
  FMD is a non-invasive technique. It was assessed using an ultrasound approach with a high-resolution linear array transducer coupled with computer-assisted analysis software. With this software, changes in the brachial artery could be assessed in real-time through an automated edge detection system. Longitudinal images of the brachial artery were obtained with the transducer fixed on the medial aspect of the dominant arm, approximately 2 cm above the medial epicondyle of the humerus. The transducer was fixed on the arm by a special arm-holding device. The brachial artery diameter was acquired as per a 30 s baseline measure, after which a cuff was placed around forearm (3 cm above wrist) and inflated to 250 mm Hg for 5 min. After cuff deflation, the brachial artery diameter was continuously monitored for 2-4 min to detect the peak artery diameter. FMD was determined as the percentage change in diameter from baseline to peak arterial diameter.
Measurement of digital volume increase by RHI (Reactive Hyperhemia Index), (Endo-PAT2000; Itamar Medical Ltd, Israel). | Visit 1: Day 0
  RHI is a non-invasive technique. It's measure with a digital plethysmography device that records pulsatile fluctuations in digital volume at rest and during reactive hyperemia. For the RH-PAT procedure, a peripheral arterial tonometry probe was placed on the right index finger and a control tonometry probe was also placed on the left index finger to eliminate sympathetic nerve effects. In the RH-PAT procedure, the RHI value was calculated as the ratio of the reactive hyperemia between the two hands.
Measurement of digital volume increase by RHI (Reactive Hyperhemia Index), (Endo-PAT2000; Itamar Medical Ltd, Israel). | Visit 3: Day 0+1 year
  RHI is a non-invasive technique. It's measure with a digital plethysmography device that records pulsatile fluctuations in digital volume at rest and during reactive hyperemia. For the RH-PAT procedure, a peripheral arterial tonometry probe was placed on the right index finger and a control tonometry probe was also placed on the left index finger to eliminate sympathetic nerve effects. In the RH-PAT procedure, the RHI value was calculated as the ratio of the reactive hyperemia between the two hands.
Microcirculation measurement by FLD (Flow Laser Doppler), PeriFlux® (Perimed) | Visit 1: Day 0
  The Flowmetry by Laser Doppler (FLD) is a non-invasive and validated technique for continuous measurement of the endothelial dependent reactivity in local microcirculation. The flow estimated by this technique is based on the assessment of the Doppler shift of low-power laser light, which is scattered by moving red blood cells. Vascular endothelial function in the micro-vascular compartment is assessed using the laser-doppler system PeriFlux 5010 (Perimed) at the level of the skin of the hands by following the response to a reactive hyperemia induced by a temporary occlusion of the brachial artery (same stimulus as for FMD measurement).
Microcirculation measurement by FLD (Flow Laser Doppler), PeriFlux® (Perimed) | Visit 3: Day 0+1 year
  The Flowmetry by Laser Doppler (FLD) is a non-invasive and validated technique for continuous measurement of the endothelial dependent reactivity in local microcirculation. The flow estimated by this technique is based on the assessment of the Doppler shift of low-power laser light, which is scattered by moving red blood cells. Vascular endothelial function in the micro-vascular compartment is assessed using the laser-doppler system PeriFlux 5010 (Perimed) at the level of the skin of the hands by following the response to a reactive hyperemia induced by a temporary occlusion of the brachial artery (same stimulus as for FMD measurement).
Sphygmocor CPV® (Atcor Medical) large artery stiffness measurement (PWV) | Visit 1: Day 0
  The carotid-femoral Pulse Wave Velocity (PWV) is an established index of arterial stiffness. Pulse, which travels at a higher velocity in stiff arterial vessels, is calculated from measurements of pulse transit time and the distance travelled between the 2 considered recording sites (i.e., carotid artery and femoral artery). The measurements are performed using a validated non-invasive device (SphygmoCor; AtCor Medical Pty. Ltd.) that allows online pulse wave recording and automatic PWV calculation [PWV = distance (m)/transit time (s)].
Sphygmocor CPV® (Atcor Medical) large artery stiffness measurement (PWV) | Visit 3: Day 0+1 year
  The carotid-femoral Pulse Wave Velocity (PWV) is an established index of arterial stiffness. Pulse, which travels at a higher velocity in stiff arterial vessels, is calculated from measurements of pulse transit time and the distance travelled between the 2 considered recording sites (i.e., carotid artery and femoral artery). The measurements are performed using a validated non-invasive device (SphygmoCor; AtCor Medical Pty. Ltd.) that allows online pulse wave recording and automatic PWV calculation [PWV = distance (m)/transit time (s)].
Evaluation of the Abdominal Aorta Calcification (AAC) (Kauppila score) | Visit 0: Day 0-1 month
  The Kauppila score is used to estimate the existence and severity of AAC. This semi-quantitative score is used to assign a score from 0 to 3, depending on the severity of vascular calcification, for the anterior and posterior walls of the aortic vessel wall, opposite each lumbar vertebrae from L1 to L4. A maximum score of 24 is thus obtained.
Evaluation of the Abdominal Aorta Calcification (AAC) (Kauppila score) | Visit 3: Day 0+1 year
  The Kauppila score is used to estimate the existence and severity of AAC. This semi-quantitative score is used to assign a score from 0 to 3, depending on the severity of vascular calcification, for the anterior and posterior walls of the aortic vessel wall, opposite each lumbar vertebrae from L1 to L4. A maximum score of 24 is thus obtained.
Strength, Assistance with walking, Rising from a chair, Climbing stairs, and Falls (SARC-F) questionnaire | Visit 1: Day 0
  Consists of 5 questions and a score higher than 4 suggests the presence of sarcopenia (or age-related muscular dystrophy). On the other hand, if the score is less than or equal to 3, the patient is diagnosed as "non-sarcopenic" but tests must be repeated regularly in clinical practice.
Strength, Assistance with walking, Rising from a chair, Climbing stairs, and Falls (SARC-F) questionnaire | Visit 3: Day 0+1 year
  Consists of 5 questions and a score higher than 4 suggests the presence of sarcopenia (or age-related muscular dystrophy). On the other hand, if the score is less than or equal to 3, the patient is diagnosed as "non-sarcopenic" but tests must be repeated regularly in clinical practice.
Short Physical Performance Battery (SPPB) Questionnaire | Visit 1: Day 0
  The Short Physical Performance Battery is the sum of the scores on three criteria: the balance test, the walking speed test and the chair lift test. This test is used to evaluate the physical performance of an individual. Adding the scores of all the tests gives an overall performance score. A score below 8 is an indicator of risk of sarcopenia (0-6 low performance 7-9, intermediate; 10-12 high).
Short Physical Performance Battery (SPPB) Questionnaire | Visit 3: Day 0+1 year
  The Short Physical Performance Battery is the sum of the scores on three criteria: the balance test, the walking speed test and the chair lift test. This test is used to evaluate the physical performance of an individual. Adding the scores of all the tests gives an overall performance score. A score below 8 is an indicator of risk of sarcopenia (0-6 low performance 7-9, intermediate; 10-12 high).
Evaluation of the muscular strength | Visit 1: Day 0
  A dynamometer measures grip strength, which decreases with age and is associated with more sarcopenia and cardiovascular comorbidities. The dynamometer is held in the dominant hand, in a sitting position, elbow bent at 90°, shoulders relaxed and forearm in a neutral position. The measurement is taken twice and the highest value is retained. Muscle strength is low when the grip strength is less than 27kg for men or 16kg for women.
Evaluation of the muscular strength | Visit 3: Day 0+1 year
  A dynamometer measures grip strength, which decreases with age and is associated with more sarcopenia and cardiovascular comorbidities. The dynamometer is held in the dominant hand, in a sitting position, elbow bent at 90°, shoulders relaxed and forearm in a neutral position. The measurement is taken twice and the highest value is retained. Muscle strength is low when the grip strength is less than 27kg for men or 16kg for women.
Body composition measurement on Dual energy X-ray Absorptiometry (DXA) | Visit 0: Day 0-1 month
  Body composition analysis by DXA, and quantification of appendicular muscle mass, is the reference method for the diagnosis of sarcopenia. It consists of measuring the appendicular skeletal mass (ASM), i.e. the muscle mass of the upper and lower limbs, or the ASM index (ASMI = ASM/height2). Sarcopenia is confirmed when the ASM is less than 20kg in men and 15kg in women or when the ASMI is less than 7kg/m2 in men and 5.5kg/m2 in women.
Body composition measurement on Dual energy X-ray Absorptiometry (DXA) | Visit 3: Day 0+1 year
  Body composition analysis by DXA, and quantification of appendicular muscle mass, is the reference method for the diagnosis of sarcopenia. It consists of measuring the appendicular skeletal mass (ASM), i.e. the muscle mass of the upper and lower limbs, or the ASM index (ASMI = ASM/height2). Sarcopenia is confirmed when the ASM is less than 20kg in men and 15kg in women or when the ASMI is less than 7kg/m2 in men and 5.5kg/m2 in women.
The Brief Pain Inventory Questionnaire (BPI) | Visit 1: Day 0
  This self-assessment scale allows the patient to characterize the pain in terms of its intensity and its psychosocial repercussions by means of 11 scales rated from 0 (no pain or does not bother) to 10 (the most horrible pain you can imagine or completely bothers you).
  The BPI also asks the patient to black out the painful areas on a diagram (front and back) and to put an "S" if the pain is on the surface or a "P" if it is deep. The questionnaire also asks the patient to indicate what treatment or medication he or she is taking for the pain and what percentage improvement has been obtained.
The Brief Pain Inventory Questionnaire (BPI) | Visit 3: Day 0+1 year
  This self-assessment scale allows the patient to characterize the pain in terms of its intensity and its psychosocial repercussions by means of 11 scales rated from 0 (no pain or does not bother) to 10 (the most horrible pain you can imagine or completely bothers you).
  The BPI also asks the patient to black out the painful areas on a diagram (front and back) and to put an "S" if the pain is on the surface or a "P" if it is deep. The questionnaire also asks the patient to indicate what treatment or medication he or she is taking for the pain and what percentage improvement has been obtained.
The Numerical Pain Scale | Visit 1: Day 0
  This scale allows the patient to rate the pain on a scale with a minimum score of 0 (no pain) and a maximum score of 10 (worst pain).
The Numerical Pain Scale | Visit 3: Day 0+1 year
  This scale allows the patient to rate the pain on a scale with a minimum score of 0 (no pain) and a maximum score of 10 (worst pain).
Measurement of the threshold of sensitivity and pain perception induced by a thermal stimulus (hot and cold) at the Pathway - Médoc®. | Visit 1: Day 0
  The measurements will be performed using an ATS thermode applied to the dominant arm of the patients. The Pathway-Medoc system associated with the thermode allows, from a base value of 32°C, to deliver adjustable temperature peaks (in the hot or in the cold and according to a regular slope of 1°C) and controlled by fast feedback, which allows to adapt to the different sensitivity thresholds of the C and A fibers. This device will be used to evaluate: the sensitivity threshold to heat, the sensitivity threshold to cold, the pain threshold to heat and the pain threshold to cold. The determination of each threshold will be established by an average of three measurements.
Measurement of the threshold of sensitivity and pain perception induced by a thermal stimulus (hot and cold) at the Pathway - Médoc®. | Visit 3: Day 0+1 year
  The measurements will be performed using an ATS thermode applied to the dominant arm of the patients. The Pathway-Medoc system associated with the thermode allows, from a base value of 32°C, to deliver adjustable temperature peaks (in the hot or in the cold and according to a regular slope of 1°C) and controlled by fast feedback, which allows to adapt to the different sensitivity thresholds of the C and A fibers. This device will be used to evaluate: the sensitivity threshold to heat, the sensitivity threshold to cold, the pain threshold to heat and the pain threshold to cold. The determination of each threshold will be established by an average of three measurements.
Central sensitization tests, measurement of the Conditioned Pain Modulation (CPM) effect | Visit 1: Day 0
  The patients are seated, the ATS thermode associated with the Pathway is applied to the dominant forearm. From the baseline value of 32°C, the Pathway delivers a "Pain 60 / Test stimulus" for 10 seconds, and the patient scores the pain on a visual numerical scale from 0 to 100. Then, the Pathway delivers a "Pain 60 / Test stimulus" for 30 seconds, and the patient scores the pain on the same scale. Fifteen minutes after the end of the two stimulations, the patient immersed the non-dominant arm for 60 seconds in a water bath at 46.5°C. Then a second identical sequence of 10 and 30 second stimulations was performed, with the scores recorded after each stimulation on the visual numerical scale from 0 to 100. The CPM effect is measured by taking the difference between the pain scores on the visual numerical scale before and after immersion.
Central sensitization tests, measurement of the Conditioned Pain Modulation (CPM) effect | Visit 3: Day 0+1 year
  The patients are seated, the ATS thermode associated with the Pathway is applied to the dominant forearm. From the baseline value of 32°C, the Pathway delivers a "Pain 60 / Test stimulus" for 10 seconds, and the patient scores the pain on a visual numerical scale from 0 to 100. Then, the Pathway delivers a "Pain 60 / Test stimulus" for 30 seconds, and the patient scores the pain on the same scale. Fifteen minutes after the end of the two stimulations, the patient immersed the non-dominant arm for 60 seconds in a water bath at 46.5°C. Then a second identical sequence of 10 and 30 second stimulations was performed, with the scores recorded after each stimulation on the visual numerical scale from 0 to 100. The CPM effect is measured by taking the difference between the pain scores on the visual numerical scale before and after immersion.
The Pittsburgh Sleep Quality Index (PSQI) | Visit 1: Day 0
  The PSQI is a self-administered questionnaire with 19 items. It was developed to measure sleep quality in the month prior to the patient interview. This questionnaire includes 7 components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, hypnotic medication use and daytime dysfunction.
  The global score (0 to 21) is obtained by adding the sub-scores of the 7 components, each ranging from 0 to 3 points. In the absence of an answer to one or more questions, the subtotal using this question cannot be calculated and will affect the overall score.
  The higher the overall score, the greater the impairment in sleep quality. An overall score >5 is an indicator of sleep disturbance.
The Pittsburgh Sleep Quality Index (PSQI) | Visit 3: Day 0+1 year
  The PSQI is a self-administered questionnaire with 19 items. It was developed to measure sleep quality in the month prior to the patient interview. This questionnaire includes 7 components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, hypnotic medication use and daytime dysfunction.
  The global score (0 to 21) is obtained by adding the sub-scores of the 7 components, each ranging from 0 to 3 points. In the absence of an answer to one or more questions, the subtotal using this question cannot be calculated and will affect the overall score.
  The higher the overall score, the greater the impairment in sleep quality. An overall score >5 is an indicator of sleep disturbance.
The 36-Item Short Form Survey (SF-36) | Visit 1: Day 0
  The quality of life of patients is assessed by the general questionnaire 36-Item Short Form Survey (SF-36) which can be administered by self or hetero-questionnaire. The SF-36 questionnaire was developed from the Medical Outcome Study, a 149-item questionnaire that was developed to assess how the American healthcare system affects the outcome of care. The SF-36 questionnaire is composed of 36 items and makes it possible to assess the physical and mental health of an individual using eleven questions relating to eight aspects of health: Physical activity, limitations due to physical state, physical pain, perceived health, vitality, life and relationship with others, limitations due to the mental state and mental health. Scores between 0 and 100 are determined. Scores tending towards 100 indicate a better quality of life.
The 36-Item Short Form Survey (SF-36) | Visit 3: Day 0+1 year
  The quality of life of patients is assessed by the general questionnaire 36-Item Short Form Survey (SF-36) which can be administered by self or hetero-questionnaire. The SF-36 questionnaire was developed from the Medical Outcome Study, a 149-item questionnaire that was developed to assess how the American healthcare system affects the outcome of care. The SF-36 questionnaire is composed of 36 items and makes it possible to assess the physical and mental health of an individual using eleven questions relating to eight aspects of health: Physical activity, limitations due to physical state, physical pain, perceived health, vitality, life and relationship with others, limitations due to the mental state and mental health. Scores between 0 and 100 are determined. Scores tending towards 100 indicate a better quality of life.
The Hospital Anxiety and Depression Scale (HAD) | Visit 1: Day 0
  It is a self-administered questionnaire completed by the patient and based on the Hamilton scale. The HAD scale is a tool for screening for anxiety and depressive disorders. It includes 14 items rated from 0 to 3. Seven questions relate to anxiety (total A) and seven others to the depressive dimension (total D), thus making it possible to obtain two scores (maximum score for each score = 21).
  To screen for anxiety and depressive symptomatology, the following interpretation can be proposed for each of the scores (A and D): ≤ 7: normal case; 8 to 10: borderline case; ≥ 11: abnormal case.
The Hospital Anxiety and Depression Scale (HAD) | Visit 3: Day 0+1 year
  It is a self-administered questionnaire completed by the patient and based on the Hamilton scale. The HAD scale is a tool for screening for anxiety and depressive disorders. It includes 14 items rated from 0 to 3. Seven questions relate to anxiety (total A) and seven others to the depressive dimension (total D), thus making it possible to obtain two scores (maximum score for each score = 21).
  To screen for anxiety and depressive symptomatology, the following interpretation can be proposed for each of the scores (A and D): ≤ 7: normal case; 8 to 10: borderline case; ≥ 11: abnormal case.
Distribution of gene polymorphisms using OpenArray technology | Visit 1: Day 0
  Blood sampling: 4 aliquots of 1 ml will be taken from the whole blood sample on EDTA tube, then frozen at -80°C in the premises of the PIC/CIC Inserm 1405, Clermont-Ferrand, France for subsequent analysis.
MicroRNA analysis using OpenArray technology will be performed on 48 patients | Visit 1: Day 0
  Genome-wide association studies highlight that genetic factors are possibly responsible of osteoporosis, and several potential candidate genes have been found to be associated to osteoporosis. The participants will be genotyped for selected SNPs (OpenArray technology) that have been previously investigated in relation to osteoporosis susceptibility, symptoms or potential mechanisms.
  Blood sampling: 1 EDTA tube of 6 ml will be collected for microRNA. The tube will then be centrifuged and 6 aliquots of 0.5 ml will be prepared (centrifugation 2500G/ 10 min/4°C) then frozen and stored at - 80°C in the premises of the PIC/CIC Inserm 1405, Clermont-Ferrand, France for subsequent analysis.
MicroRNA analysis using OpenArray technology will be performed on 48 patients | Visit 3: Day 0+1 year
  Genome-wide association studies highlight that genetic factors are possibly responsible of osteoporosis, and several potential candidate genes have been found to be associated to osteoporosis. The participants will be genotyped for selected SNPs (OpenArray technology) that have been previously investigated in relation to osteoporosis susceptibility, symptoms or potential mechanisms.
  Blood sampling: 1 EDTA tube of 6 ml will be collected for microRNA. The tube will then be centrifuged and 6 aliquots of 0.5 ml will be prepared (centrifugation 2500G/ 10 min/4°C) then frozen and stored at - 80°C in the premises of the PIC/CIC Inserm 1405, Clermont-Ferrand, France for subsequent analysis.
Study of the microbiota will be performed on 48 patients | Visit 1: Day 0
  Identification of bacterial biodiversity by a genetic sequencing analysis of bacterial DNA. The patient must collect the stool by following the technical instructions described in the explanatory leaflet that will be provided. She must then respect the procedure for the conservation and transport of the stool described in this document. The samples will be stored and frozen at -80°C at the PIC/ CIC Inserm 1405, Clermont-Ferrand, France until subsequent analysis.
Study of the microbiota will be performed on 48 patients | Visit 3: Day 0+1 year
  Identification of bacterial biodiversity by a genetic sequencing analysis of bacterial DNA. The patient must collect the stool by following the technical instructions described in the explanatory leaflet that will be provided. She must then respect the procedure for the conservation and transport of the stool described in this document. The samples will be stored and frozen at -80°C at the PIC/ CIC Inserm 1405, Clermont-Ferrand, France until subsequent analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Eva PICKERING, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU clermont-ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Pickering ME, Morel V, Nicolas M, Duale C, Sortais E, Graven-Nielsen T, Pereira B, Pickering G. Quantitative sensory testing of pain in osteoporosis: a pilot randomized clinical trial with magnesium supplementation. Aging Clin Exp Res. 2026 Jan 21. doi: 10.1007/s40520-025-03317-9. Online ahead of print. PMID 41566091